CLINICAL TRIAL: NCT02922777
Title: Phase 1 Trial of Dose Escalated BGB324 in Combination With Docetaxel for Previously Treated Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Trial of Dose Escalated BGB324 in Previously Treated Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Tech University Health Sciences Center (Other); BerGenBio ASA (Industry)
Responsible Party: Principal Investigator, David E Gerber, Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052015-077
Record Dates: First submitted 2016-05-19; First posted 2016-10-04 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bemcentinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BGB324 in combination with docetaxel (Experimental): The dose of docetaxel will be 75 mg/m2 given IV every 21 days. The dose of BGB324 will be escalated in a standard 3+3 fashion until a maximum tolerated dose is determined.
  Interventions: Drug: BGB324; Drug: Docetaxel

INTERVENTIONS:
Drug: BGB324 — 75 mg/m2 every 21 days
Drug: Docetaxel — 75 mg/m2 given IV every 21 days
  Other Names: Taxotere

SUMMARY:
This study is being done to evaluate the safety of the investigational study drug, BGB324 when administered in combination with docetaxel, and to establish the maximum tolerated dose.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related deaths worldwide with an estimated incidence of 1.6 million cases resulting in 1.4 million deaths in annually. Non-small-cell lung cancer (NSCLC) represents 80-85% of cases, and adenocarcinoma is the most common histology.2 The majority of NSCLC patients present with advanced or metastatic disease that is not amenable to surgical resection. Platinum-based combination chemotherapy has reached a therapeutic plateau with a median overall survival (OS) of 7.4 to 9.9 months.

BGB324 is a potent selective small molecule inhibitor of Axl, a surface membrane protein kinase receptor that is over-expressed in many metastatic solid tumors and has been identified as a marker of a poor prognosis in patients with non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for the study if the following criteria are met:

1. Provision of written informed consent to participate in this investigational study
2. Histologically or cytologically confirmed advanced (stage 4, according to the American Joint Committee on Cancer [AJCC] Staging manual) NSCLC
3. Up to three previous lines of therapy, of which one must have been a platinum-based doublet therapy and no more than two were cytotoxic chemotherapy.
4. Radiographic disease recurrence or progression during or after the last line of chemotherapy
5. Patients with known activating EGFR mutations or ALK rearrangements should have progressed after appropriate targeted treatment in addition to progressing during or after platinum-based doublet chemotherapy
6. European Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Age 18 years or older
8. Measurable or evaluable disease according to RECIST v1.1
9. Previously treated brain metastases (surgery and/or radiation therapy) are eligible, provided that patients are asymptomatic and not requiring corticosteroids
10. The following minimum intervals are required between prior treatment and initiation of study therapy:

    Cytotoxic chemotherapy: 3 weeks Molecularly targeted therapy or immunotherapy: 2 weeks Conventional fractionated radiation therapy: 2 weeks Stereotactic radiation therapy: 1 week Major surgery: 3 weeks
11. Adequate hematologic function (absolute neutrophil count [ANC] ≥ 1500 cells/µL; hemoglobin ≥ 9 g/dL; platelets ≥ 100,000/µL
12. Adequate renal function (serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation)
13. Adequate hepatic function: total bilirubin ≤ upper limit of normal [ULN], alanine aminotransferase [ALT] ≤ 1.5 x ULN, aspartate aminotransferase [AST] ≤ 1.5 x ULN). ALT and AST ≤ 5x ULN if documented liver metastases
14. Previous treatment-associated toxicities resolved to CTCAE grade ≤2 (except alopecia)
15. Adequate archival tissue (10-15 slides, or 5 slides with 3 sections per slide) for biomarker analysis
16. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to taking their first dose of BGB324. Male patients and female patients of reproductive potential must agree to practice highly effective methods of contraception (such as hormonal implants, combined oral contraceptives, injectable contraceptives, intrauterine device with hormone spirals, total sexual abstinence, vasectomy) throughout the study and for ≥3 months after the last dose of BGB324. Female patients are considered NOT of childbearing potential if they have a history of surgical sterility, including tubal ligation, or evidence of post-menopausal status defined as any of the following:

    * Natural menopause with last menses >1 year ago
    * Radiation induced oophorectomy with last menses >1 year ago
    * Chemotherapy induced menopause with last menses >1 year ago

Exclusion Criteria

A patient is excluded from the study if any of the following criteria are met:

1. Pregnant or lactating
2. Abnormal left ventricular ejection fraction on echocardiography (less than the lower limit of normal for a patient of that age at the treating institution or <45%)
3. History of an ischemic cardiac event including myocardial infarction within 3 months of study entry
4. NSCLC with evidence of a centrally cavitating lesion
5. Peripheral neuropathy NCI CTCAE ≥Grade 2 at baseline
6. Pulmonary hemorrhage or hemoptysis > 2.5 mL blood within 6 weeks (or within 2 weeks if source definitively treated [eg, radiation therapy or bronchoscopic procedure])
7. Congestive cardiac failure of >Grade 2 severity according to the NYHA defined as symptomatic at less than ordinary levels of activity
8. Unstable cardiac disease, including unstable angina or unstable hypertension, as defined by the need for change in medication for lack of disease control within the last three months
9. History or presence of sustained bradycardia (less than or equal to 60 BPM) or history of symptomatic bradycardia, left bundle branch block, cardiac pacemaker or significant atrial tachyarrhythmias , as defined by the need for treatment
10. Previous treatment with docetaxel or an Axl inhibitor
11. Current treatment with agents that may prolong QT interval and may cause Torsade de Points which cannot be discontinued at least five half-lives prior to treatment. Please see Appendix J for list of relevant medications
12. Known family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy
13. Previous history of Grade 3 or worse drug-induced QTc prolongation requiring treatment withdrawal
14. Screening 12-lead ECG with a measurable QTc interval according to Fridericia's correction >450 ms
15. Ongoing infection requiring systemic treatment
16. Inability to tolerate oral medication
17. Impaired coagulation as evidenced by:

    * INR >1.5 times ULN, or
    * aPTT > 1.5 times ULN
18. Clinically active existing gastrointestinal disease affecting drug absorption, such as celiac disease or Crohn's disease
19. Previous bowel resection anticipated to affect drug absorption
20. Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
21. Treatment with any medication which is predominantly metabolized by CYP3A4 and has a narrow therapeutic index
22. Active, uncontrolled central nervous system (CNS) disease
23. Known active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses (screening not required)
24. Major surgery within 28 days prior to the start of BGB324, excluding skin biopsies and procedures for insertion of central venous access devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of BGB324 in combination with docetaxel | 42 days or 2 cycles of 21 days
  Determine and recommended the Phase 2 dose of BGB324 administered with the standard dose of docetaxel in patients in NSCLC by pharmacodynamics and pharmacokinetic assessments.

CONTACTS AND LOCATIONS:
Overall Officials: David E Gerber, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Covenant Health Systems/Joe Arrington Cancer Treatment and Research Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02922777/Prot_SAP_000.pdf